CLINICAL TRIAL: NCT00681187
Title: A Phase IV, International, Open-label, Randomised, Cross-over Study to Assess Patient Preference and Health Economy in Patients With Neuroendocrine Tumours, Treated With Lanreotide Autogel Given as Self Administration.
Brief Title: Somatuline Autogel Preference and Health Economy Study
Acronym: SAPHE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A-99-52030-216; 2007-006514-42 (EudraCT Number)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Neuroendocrine Tumour With Carcinoid Symptoms
MeSH Terms: interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — 90 mg or 120 mg once every 28th day

SUMMARY:
The primary aim of this study is to assess which method of lanreotide Autogel administration patients with neuroendocrine tumours prefer - self/partner administrations or healthcare provided administrations. The study will also assess if self/partner administration can be performed without loss of efficacy and with a preserved safety profile. The impact of self/partner administration on resource utilisation and costs will be studied. In addition, we will also assess the healthcare provider's experience of the two administration practices.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent from the patient and their partner (if the partner will be administering the lanreotide Autogel injections during the self administration period)
* Male or female aged 18 years of age or older
* Treated with lanreotide Autogel 90 or 120 mg every 28th day for carcinoid symptoms on a stable dose for at least 3 months prior to inclusion. The patient is presumed to be clinically stable during the coming months
* Neuroendocrine tumour confirmed by biopsy and visible on radiology

Exclusion Criteria:

* Has a history of hypersensitivity to the Investigational Medicinal Product or drugs with a similar chemical structure
* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study
* Has a life expectancy less than a year, as judged by the Investigator
* The patient or their partner is not considered competent in injection technique, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- Denmark (2):
  - Aarhus University Hospital / Medisinsk afd. V, Aarhus
  - Odense Univeristy Hospital / S-AMB, Odense
- Norway (3):
  - Haukeland University Hospital / Kreftafd, Bergen
  - University Hospital North-Norway / GastroLab, Tromsø
  - S:t Olavs Hospital / Medisinsk Afd, Trondheim
- Sweden (5):
  - Sahlgrenska University Hospital / Kirurgkliniken, Gothenburg
  - Linköping University Hospital / Onkologen, Linköping
  - Karolinska University Hospital, Huddinge / GastroCentrum Medicin, Stockholm
  - Karolinska University Hospital, Solna / Kirurgmottagningen, Stockholm
  - Akademiska Hospital/ Kliniken f onkologisk endokrinologi, Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from ninety-four subjects was reviewed in hospital clinics in Denmark, Norway and Sweden. Of which 32 were ineligible, 36 were eligible but chose not to participate due to lack of motivation, satisfaction with current form of administration or fear of self-injection and 26 were included. Patients were recruited from Jun-08 to Jan-10.
Groups:
- Group 1 Self or Partner First Then HCP Administration: Started with a training period where the subject or partner performed two or three training injections under supervision of a Healthcare Professional (HCP) at a healthcare provider facility. The training injections were followed by a self administration block of three subsequent unsupervised injections every 28th day at the subject's home. A healthcare administration block followed the self administration block with three HCP provided injections according to clinical routine every 28th day.
- Group 2 HCP Then Self or Partner Administration: Started with a healthcare administration block with three HCP provided injections according to clinical routine every 28th day. A training period followed the healthcare administration block with two or three training injections performed by the subject or partner under supervision at the healthcare provider facilities. A self-administration block followed the training injections with 3 subsequent unsupervised injections every 28th day at the subject's home. The subject visited the clinic for a follow-up visit 14 days after the last self-partner administered injection.
Period: Overall Study
Arm/Group | Group 1 Self or Partner First Then HCP Administration | Group 2 HCP Then Self or Partner Administration
Started | 11 | 15
Completed | 10 | 13
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Self or Partner First Then HCP Administration: Self or partner administration followed by HCP administration.
- Group 2 HCP Then Self or Partner Administration: Administration by HCP then self or partner administration.
- Total: Total of all reporting groups
Arm/Group | Group 1 Self or Partner First Then HCP Administration | Group 2 HCP Then Self or Partner Administration | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.5) | 60.0 (12.7) | 61.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Denmark | 3 | 4 | 7
  Norway | 1 | 3 | 4
  Sweden | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Subject Preference for Self or Partner Administration
Description: A global question was asked: 'If you could choose, which administration method would you like to use on a regular basis?' A) Healthcare professional provided injection B) Self/ partner administered injection
Time Frame: Between week 30 to 34
Population: Analysis was performed on Intention to Treat population defined as all randomised subjects with ≥ 1 dose of study medication and with a preference assessment recorded
Measure: Number; unit: participants
Arm/Group | Group 1 Self or Partner First Then HCP Administration | Group 2 HCP Then Self or Partner Administration
Number analyzed (Participants) | 11 | 14
participants | 10 [58.7 to 99.8] | 12 [57.2 to 98.2]

2. Secondary Outcome: Number of Patients Stating at Least One Injection Interfered With Daily Activities
Description: The subject was asked: 'Does the treatment administration used today interfere with your daily activities?'
Time Frame: Between baseline to week 32, after each injection (8-9 injections)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Training Period: The training period was where the subject or partner performed two or three training injections under supervision of a HCP at a healthcare provider facility.
- Self or Partner Administration: The self or partner administration block (after training period) included three unsupervised injections every 28th day at the subject's home.
- HCP Administration: A healthcare administration block included three HCP provided injections according to clinical routine every 28th day at the healthcare provider facility.
Arm/Group | Training Period | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 25 | 25 | 25
Participants | 6 | 2 | 6

3. Secondary Outcome: Number of Patients Stating at Least One Injection Negatively Interfered With Psychological Wellbeing
Description: The subject was asked: 'Does the treatment administration used today negatively interfere with your psychological wellbeing?'
Time Frame: Between baseline to week 32, after each injection (8-9 injections)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Training Period | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 25 | 25 | 25
participants | 4 | 2 | 1

4. Secondary Outcome: Days Sick Leave
Description: Health care and patient costs associated with the treatment of carcinoid symptoms in subjects treated with lanreotide Autogel were assessed through recording loss of production for subject through total number of days sick leave of the employed patients (n=6).
Time Frame: Group 1 - between week 8 to 20 (self or partner administration), between week 20 to 32 (HCP administration). Group 2 - between week 20 to 32 (self or partner administration), between week 0 to week 12 (HCP administration)
Population: Safety population: all randomised subjects with at least one dose of study medication. Two of the six subjects reported sick leave during the study. One subject was absent for one day due to unknown reason, the other was absent for 22 days due to surgery of metastasis.
Measure: Number; unit: days
Groups:
- Self or Partner Administration: The self or partner administration block (after the training period) included three unsupervised injections every 28th day at the subject's home.
Arm/Group | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 6 | 6
days | 23 | 0

5. Secondary Outcome: Total Number of Visits to HCP Due to Carcinoid Symptoms
Description: Health care and patient costs associated with the treatment of carcinoid symptoms in subjects treated with lanreotide Autogel were assessed by recording the total number of visits made by participants (n=12) to HCP due to carcinoid symptoms.
Time Frame: as for outcome 4
Population: Safety population: all randomised subjects with at least one dose of study medication
Measure: Number; unit: visits
Groups:
- Self or Partner Administration: The self or partner administration block (after the training) included three unsupervised injections every 28th day at the subject's home.
Arm/Group | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 12 | 12
visits | 17 | 25

6. Secondary Outcome: Perceived Symptom Control Evaluation in Respect to Episodes of Flushing
Description: Participants were asked how they perceived the symptoms in respect to episodes of flushing since the last injection. Participants included in the study were previously treated with lanreotide Autogel and therefore the assessment at baseline was made in comparison to their previous injection outside of the study protocol.
Time Frame: Group 1 - baseline, week 16 to 20 (self or partner administration) and week 30 to 34 (HCP administration). Group 2 - baseline, week 12 (HCP administration) and week 30 (self or partner administration).
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Baseline: Baseline refers to the last non-study visit at the clinic.
Arm/Group | Baseline | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 25 | 25 | 25
participants
  Worsened | 0 | 1 | 1
  Similar | 24 | 21 | 20
  Improved | 1 | 2 | 4
  Missing | 0 | 1 | 0

7. Secondary Outcome: Perceived Symptom Control Evaluation in Respect to Episodes of Diarrhoea
Description: Participants were asked how they perceived the symptoms in respect to episodes of diarrhoea since the last injection. Participants included in the study were previously treated with lanreotide autogel and therefore the assessment at baseline was made in comparison to previous injection outside of the study protocol.
Time Frame: Group 1 - baseline, week 16 to 20 (self or partner administration) and week 30 to 34 (HCP administration). Group 2 - baseline, week 12 to 16 (HCP administration) and week 30 to 34 (self or partner administration).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Baseline | Self or Partner Administration | HCP Administration
Number analyzed (Participants) | 25 | 25 | 25
participants
  Worsened | 1 | 4 | 0
  Similar | 22 | 17 | 24
  Improved | 2 | 3 | 1
  Missing | 0 | 1 | 0

8. Secondary Outcome: Chromogranin A Levels
Description: Biochemical control was assessed by analysing chromogranin A levels at each site visit, which was mandatory for all subjects.
  'Before self or partner administration' was assessed at baseline for group 1 and at week 12 for group 2.
  'After self or partner administration' was assessed at week 16 to 20 for group 1 and at week 12 for group 2.
  'Before HCP administration' was assessed at week 16 to 20 for group 1 and at baseline for group 2.
  'After HCP administration' was assessed at week 30 to 34 for group 1 and week 12 for group 2.
Time Frame: Group 1 - Baseline, week 16 to 20 and 30 to 34. Group 2 - Baseline, week 12 and 30 to 34.
Population: ITT population that had hormone levels assessed at each administration block.
Measure: Mean (Standard Deviation); unit: nmol/l
Groups:
- Before Self or Partner Administration: Before self or partner administration block (after training period) which included three unsupervised injections every 28th day at the subject's home.
- After Self or Partner Administration: After the self or partner administration block which included three unsupervised injections every 28th day at the subject's home.
- Before HCP Administration: Before the healthcare administration block which included three HCP provided injections according to clinical routine every 28th day at the healthcare provider facility.
- After HCP Administration: After the healthcare administration block which included three HCP provided injections according to clinical routine every 28th day at the healthcare provider facility.
Arm/Group | Before Self or Partner Administration | After Self or Partner Administration | Before HCP Administration | After HCP Administration
Number analyzed (Participants) | 22 | 22 | 22 | 22
nmol/l | 37.48 (58.35) [11.61 to 63.35] | 47.85 (74.89) [14.65 to 81.05] | 42.05 (70.74) [10.69 to 73.41] | 37.42 (57.96) [11.72 to 63.11]

9. Secondary Outcome: 5-hydroxyindoleacetic Acid (5-HIAA) Levels
Description: Biochemical control was assessed by analysing 5-HIAA levels at each site visit, which was judged as necessary by the investigator at each site.
  'Before self or partner administration' was assessed at baseline for group 1 and at week 12 for group 2.
  'After self or partner administration' was assessed at week 16 to 20 for group 1 and at week 12 for group 2.
  'Before HCP administration' was assessed at week 16 to 20 for group 1 and at baseline for group 2.
  'After HCP administration' was assessed at week 30 to 34 for group 1 and week 12 for group 2.
Time Frame: Group 1 - Baseline, week 16 to 20 and 30 to 34. Group 2 - Baseline, week 12 and 30 to 34.
Population: 5-HIAA were assessed as judged necessary by the investigator at each site.
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Before Self or Partner Administration | After Self or Partner Administration | Before HCP Administration | After HCP Administration
Number analyzed (Participants) | 12 | 12 | 12 | 12
nmol/l | 220.17 (238.32) [68.75 to 371.59] | 219.17 (227.64) [74.53 to 363.80] | 217.08 (244.32) [61.85 to 372.32] | 219.58 (218.51) [80.75 to 358.42]

10. Secondary Outcome: Healthcare Professionals With Positive Response to Specified Questions on Self or Partner Administration Method
Description: Assessed by the number of HCP with a positive response 'yes' to two questions:
  1. Based on your experience during this trial, did you feel confident in the safety of your patients?
  2. Based on your experience during this trial, would you recommend suitable patients to try self or partner administration?
Time Frame: Between week 30 to 34
Population: One HCP from each site who enrolled participants replied to the question
Measure: Number; unit: participants
Groups:
- Overall Study Group: One HCP from each site who enrolled participants answered the questions
Arm/Group | Overall Study Group
Number analyzed (Participants) | 9
participants | 9 [66.4 to 100.0]

ADVERSE EVENTS:
Arm/Group | Training Period | Self or Partner Administration | HCP Administration
Serious Adverse Events (participants affected / at risk) | 4/26 | 4/26 | 3/26
Other Adverse Events (participants affected / at risk) | 7/26 | 4/26 | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Training Period (N=26) | Self or Partner Administration (N=26) | HCP Administration (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritoneal cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Training Period (N=26) | Self or Partner Administration (N=26) | HCP Administration (N=26)
Disease progression (General disorders) | 0 (0) | 1 (2) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 1 (3) | 3 (6)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days